CLINICAL TRIAL: NCT00481858
Title: A CLL Research Consortium (CRC) Phase II Study of Kinetic Biomarker for Chronic Lymphocytic Leukemia (CLL) Prognosis
Brief Title: Kinetic Biomarker for Chronic Lymphocytic Leukemia Prognosis
Acronym: CRC011
Status: Completed | Type: Observational
Sponsor: KineMed (Industry)
Collaborators: Chronic Lymphocytic Leukemia Research Consortium (Network)
Responsible Party: Gregory Hayes, Director - Oncology, KineMed
Other Study IDs: CRC011; NCI 5R44CA097686-05
Record Dates: First submitted 2007-05-31; First posted 2007-06-04 (Estimated); Last update posted 2011-02-28 (Estimated); Status verified 2011-02

CONDITIONS: Chronic Lymphocytic Leukemia
Keywords: chronic lymphocytic leukemia; biomarker; prognosis; apoptosis; neoplasm/cancer diagnosis; stable isotope; diagnosis evaluation; outcomes; CD19; CD5
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Neoplasms

STUDY DESIGN:
Observational Model: Cohort
Biospecimen Retention: Samples With DNA — CLL cells
Oversight: Data Monitoring Committee: No

SUMMARY:
This project will attempt to validate the utilization of a stable isotope kinetic biomarker (KineMarkerTM) as a predictive test for disease progression in early stage chronic lymphocytic leukemia (CLL).

DETAILED DESCRIPTION:
Chronic Lymphocytic Leukemia (CLL), the most common leukemia in the western world, is characterized by a pathological expansion of leukemic B cells. The clinical course of CLL is remarkably heterogeneous; some patients have relatively aggressive disease requiring early treatment, others have highly indolent disease that does not require current anti-leukemia therapy until many years after diagnosis. Current staging systems have not been able to predict which patients in early or intermediate risk stages will undergo disease progression and which will undergo an indolent course. Universal treatment of all patients with early stage disease has been shown to be more harmful than beneficial. As such, early identification of patients who will have more aggressive disease soon after diagnosis has been a major goal in CLL research.

In response to this need for a reliable prognostic marker, KineMed is investigating the use of CLL kinetics as a biomarker for subsequent disease progression. This test assesses B-Cell kinetics directly through an in vivo kinetic measurement of tumor DNA synthesis and catabolism by combining 2H2O labeling and state of the art analytic instrumentation.

ELIGIBILITY:
Inclusion Criteria:

* >18 years of age
* clinical diagnosis of chronic lymphocytic leukemia
* diagnosis within previous 3 years
* Stage 0, I, or II disease
* willingness and capacity to give informed consent

Exclusion Criteria:

* current or prior cll treatment
* serious co-morbid medical condition
* patient likely to need treatment in the next 16 weeks
* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: CLL patients
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2005-07; Primary Completion 2010-07 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Hayes, Ph.D., Principal Investigator — KineMed Inc.
Locations (5):
- United States (5):
  - UCSD Medical Center, San Diego, California
  - Mayo Clinic, Rochester, Minnesota
  - North Shore-Long Island Jewish Medical Center, New Hyde Park, New York
  - Ohio State University, Columbus, Ohio
  - M.D. Anderson Cancer Center, Houston, Texas

REFERENCES:
- [Result] Messmer BT, Messmer D, Allen SL, Kolitz JE, Kudalkar P, Cesar D, Murphy EJ, Koduru P, Ferrarini M, Zupo S, Cutrona G, Damle RN, Wasil T, Rai KR, Hellerstein MK, Chiorazzi N. In vivo measurements document the dynamic cellular kinetics of chronic lymphocytic leukemia B cells. J Clin Invest. 2005 Mar;115(3):755-64. doi: 10.1172/JCI23409. PMID 15711642
- [Derived] Hayes GM, Busch R, Voogt J, Siah IM, Gee TA, Hellerstein MK, Chiorazzi N, Rai KR, Murphy EJ. Isolation of malignant B cells from patients with chronic lymphocytic leukemia (CLL) for analysis of cell proliferation: validation of a simplified method suitable for multi-center clinical studies. Leuk Res. 2010 Jun;34(6):809-15. doi: 10.1016/j.leukres.2009.09.032. Epub 2009 Oct 24. PMID 19854509
- See also: Related Info — http://www.kinemed.com